CLINICAL TRIAL: NCT00425776
Title: Treatment of Hot Flushes in Breast Cancer Patients With Acupuncture
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: K07-01
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Breast Cancer; Postmenopause
Keywords: Breast cancer; Acupuncture; Post-menopausal hot flushes; Se-estradiol; Se-endorphine
MeSH Terms: conditions — Breast Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Real acupuncture (Active Comparator)
  Interventions: Device: acupuncture
- Sham acupuncture (Sham Comparator)
  Interventions: Device: Sham acupuncture
- No intervention (No Intervention)

INTERVENTIONS:
Device: acupuncture
  Other Names: Acupuncture, hot flushes
  Arms: Real acupuncture
Device: Sham acupuncture
  Arms: Sham acupuncture

SUMMARY:
In a randomized 3-group clinical study acupuncture is used for the relief of menopausal hot flushes and sleep disturbances in women treated for breastcancer.

The three groups consists of 35 women given acupuncture once a week five times and 35 women given shamacupuncture once a week five times and 35 women with no kind of treatment. Se-estradiol and endorphin is measured before and after the acupuncture.

We want to state that acupuncture given five times once a week has a significant better effect on hot flushes and sleeping disturbances than shamacupuncture or no treatment at all.

We also want to measure if there are any changes in se-estradiol and endorphine

DETAILED DESCRIPTION:
Breast cancer patients often have a higher prevalance of menopausal symptoms with hor flushes and sleeping disturbances than women in the general population, and hormone replacement therapy is not considered suitable for breast cancer patients because an increase in oestrogen is contraindicated.

There has been some evidence that acupuncture is suitable treatment for hot flushes and therefore we had a small pilotproject where 25 women treated for breast cancer were given a course of classical body acupuncture with one 15 min treatment session per week for 5 weeks. The effekt was remarkable.

We want to prove if this effekt is significantly better than shamacupuncture or to no treatment at all.

This is a prospective, randomized and doubbleblinded study:

35 women get classical body acupuncture once a week 5 times 35 women get shamacupuncture once a week 5 times 35 women get no acupuncture. Se-estradiol and se-endorphine will be measure before start of the first acupuncture and after the first and fifth acupuncture. The women with no treatment will have blodsamples too in the beginning and at the end of the fifth week.

ELIGIBILITY:
Inclusion Criteria:

* Women older than 35 years treated for breastcancer having hot flushes and sleeping disturbances.It is not allowed to take estrogen as tablets or plaster.

Exclusion Criteria:

* Failing to give consent
* Any use of estrogen as tablets or plaster

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2007-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
using a hot flushes rating scale. | 12 weeks
Sleep disturbances yes or no | 12 weeks

SECONDARY OUTCOMES:
Measuring se-estrogen and se-endorhine before and after acupuncture | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Claus Bisgaard, Consultant, Principal Investigator — Vejle Hospital
Locations (1):
- Vejle Hospital, Vejle, Kabbeltoft 25, Denmark

REFERENCES:
- [Derived] Bokmand S, Flyger H. Acupuncture relieves menopausal discomfort in breast cancer patients: a prospective, double blinded, randomized study. Breast. 2013 Jun;22(3):320-3. doi: 10.1016/j.breast.2012.07.015. Epub 2012 Aug 18. PMID 22906948